CLINICAL TRIAL: NCT00651222
Title: Influence of Androgen Suppression Therapy for Prostate Cancer on the Timing and Onset of Fatal Myocardial Infarctions in Men Undergoing Prostate Brachytherapy
Brief Title: Influence of Hormone Therapy on Heart Attack Incidence in Men Undergoing Prostate Brachytherapy
Status: Completed | Type: Observational
Sponsor: Prostate Cancer Foundation of Chicago (Other)
Responsible Party: Brian J. Moran, MD, Prostate Cancer Foundation of Chicago
Other Study IDs: MI-PB
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Prostate Cancer; Cardiovascular Death
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All deceased patients who underwent brachytherapy at Chicago Prostate Center between 10/14/1997 and 6/15/2007
  Interventions: Other: No intervention was required

INTERVENTIONS:
Other: No intervention was required — Death records were reviewed, therefore, there was no intervention
  Other Names: Death records were reviewed, therefore, there was no intervention

SUMMARY:
The purpose of this study is to review cause of death in patients undergoing prostate brachytherapy at a single institution. Furthermore, we are analyzing patients undergoing androgen deprivation therapy and whether or not this contributed to cardiovascular deaths, specifically myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Deceased anytime after prostate brachytherapy treatment

Exclusion Criteria:

* Patients whose cause of death was unable to be determined

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients treated with prostate brachytherapy at an ambulatory surgery center
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago Prostate Center, Westmont, Illinois, United States